CLINICAL TRIAL: NCT02954029
Title: Hemostasis Pad Using Chitosan After Invasive Percutaneous Procedures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Si-Hyuck Kang, professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ezClot1
Record Dates: First submitted 2016-07-12; First posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Artery Disease; Puncture
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Study group (transradial cohort) (Experimental): device-assisted compression with ezClot pad
  Interventions: Device: ezClot (hemostasis pad); Device: Rotary compression device
- Study group (transfemoral cohort) (Experimental): manual compression with ezClot pad
  Interventions: Device: ezClot (hemostasis pad)
- Control group (transradial cohort) (Active Comparator): Rotary compression device
  Interventions: Device: Rotary compression device
- Control group (transfemoral cohort) (Active Comparator): manual compression with BloodSTOP ix pad
  Interventions: Device: BloodSTOP ix pad

INTERVENTIONS:
Device: ezClot (hemostasis pad) — ezClot pad uses chitosan, a deacetylated complex carbohydrate derived from the naturally occurring substance chitin, to accelerate blood clotting.
  Arms: Study group (transfemoral cohort); Study group (transradial cohort)
Device: BloodSTOP ix pad — BloodSTOP® pad is an etherized and oxidized regenerated cellulose matrix that achieves hemostasis by activating the intrinsic coagulation pathway.
  Arms: Control group (transfemoral cohort)
Device: Rotary compression device — Rotary compression device consists of a plastic arch and a rotary screw to deliver local pressure by moving the silicone compression pad.
  Arms: Control group (transradial cohort); Study group (transradial cohort)

SUMMARY:
Arterial access is the key step during the endovascular treatment of cardiovascular diseases. This study was designed to confirm the safety and efficacy of the hemostasis pad using chitosan in patients undergoing percutaneous procedures with arterial approach. Two cohorts will be included in this study: transradial and transfemoral cohort. Among the transfemoral cohort, the safety and efficacy of the ezClot pad will be compared with the BloodSTOP® pad (LifeScience PLUS, Palo Alto, CA, USA). The BloodSTOP® pad is an etherized and oxidized regenerated cellulose matrix that achieves hemostasis by activating the intrinsic coagulation pathway. The hypothesis will be tested among the transradial cohort that the combined use of a hemostasis pad and a compression device is superior to that of a compression device only in terms of hemostasis in patients who underwent tranradial coronary procedures.

DETAILED DESCRIPTION:
Arterial access is the key step during the endovascular treatment of cardiovascular diseases. However, failure in hemostasis of the arterial access sites is associated with high risk of complications such as bleeding, pseudoaneurysm, and arteriovenous fistula. Major bleeding events after percutaneous coronary intervention has been shown be associated with poor short-term as well as long-term prognosis. Thus, there have been a variety of approaches to quickly and effectively achieve hemostasis of the puncture site. The traditional method was to apply manual compression followed by simple dressing directly on the puncture site. Despite a long history and economic advantage, this method required prolonged hemostasis time, substantial efforts by trained practitioner, and patients' discomfort.

Use of hemostasis pad that accelerates blood clotting has become an effective alternative. The ezClot pad is a new product that uses chitosan, a deacetylated complex carbohydrate derived from the naturally occurring substance chitin. The positively charged chitosan molecules attract the negatively charged blood cells and platelets, thus promoting clots. The ability to hemostasis of chitosan has been proven with the HemCon® pad (HemCon Medical Technologies, Inc., Portland, OR, USA). This study was designed to confirm the safety and efficacy of the ezClot pad in patients undergoing percutaneous procedures with arterial approach. Two cohorts will be included in this study: transradial and transfemoral cohort. Among the transfemoral cohort, the safety and efficacy of the ezClot pad will be compared with the BloodSTOP® pad (LifeScience PLUS, Palo Alto, CA, USA). The BloodSTOP® pad is an etherized and oxidized regenerated cellulose matrix that achieves hemostasis by activating the intrinsic coagulation pathway.

Transradial approach is increasing used during coronary procedures. The most important benefit of transradial approach compared to transfemoral approach is low risk of major bleeding. Widely used method for hemostasis of radial puncture sites were manual or device-assisted compression. There is yet only a limited data regarding the use of hemostasis pad after transradial approach. The hypothesis will be tested in the transradial cohort that the combined use of a hemostasis pad and a compression device is superior to that of a compression device only in terms of hemostasis in patients who underwent transradial coronary procedures.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* patients undergoing invasive procedures via the radial or femoral arteries

Exclusion Criteria:

* congenital or acquired bleeding tendency
* platelet count <50,000/ μL
* hypersensitivity to shrimps, lobsters or beetles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Time to hemostasis | Immediately after invasive procedures

SECONDARY OUTCOMES:
Bleeding | within 24 hours
  TIMI major/minor bleeding within 24 hours
Hematoma | within 24 hours
  Hematoma within 24 hours
Retroperitoneal hematoma | within 24 hours
  Retroperitoneal hematoma within 24 hours
Pseudoaneurysm | within 24 hours
  Pseudoaneurysm within 24 hours
Vessel occlusion | within 24 hours
  Vessel occlusion within 24 hours (either 1 or 2)
  1. no palpable pulse
  2. no flow on Doppler
Dissection | within 24 hours
  Dissection of access vessel within 24 hours (either 1 or 2)
  1. observed on angiography
  2. symptomatic compromising distal flow
Surgical repair | within 24 hours
  Surgical repair within 24 hours
Vasovagal reaction | within 24 hours
  Vasovagal reaction (grade 3-4) within 24 hours

OTHER OUTCOMES:
Hb at discharge | within 24 hours
  hemoglobin (g/dL) within 24 hours
Hb at 1-month F/U | 1 month after discharge
  hemoglobin (g/dL) at 1-month outpatient follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suh JW, Mehran R, Claessen BE, Xu K, Baber U, Dangas G, Parise H, Lansky AJ, Witzenbichler B, Grines CL, Guagliumi G, Kornowski R, Wohrle J, Dudek D, Weisz G, Stone GW. Impact of in-hospital major bleeding on late clinical outcomes after primary percutaneous coronary intervention in acute myocardial infarction the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) trial. J Am Coll Cardiol. 2011 Oct 18;58(17):1750-6. doi: 10.1016/j.jacc.2011.07.021. PMID 21996385
- [Background] Eikelboom JW, Mehta SR, Anand SS, Xie C, Fox KA, Yusuf S. Adverse impact of bleeding on prognosis in patients with acute coronary syndromes. Circulation. 2006 Aug 22;114(8):774-82. doi: 10.1161/CIRCULATIONAHA.106.612812. Epub 2006 Aug 14. PMID 16908769
- [Background] Pusateri AE, Holcomb JB, Kheirabadi BS, Alam HB, Wade CE, Ryan KL. Making sense of the preclinical literature on advanced hemostatic products. J Trauma. 2006 Mar;60(3):674-82. doi: 10.1097/01.ta.0000196672.47783.fd. PMID 16531876
- [Background] Arbel J, Rozenbaum E, Reges O, Neuman Y, Levi A, Erel J, Haskia AR, Caneti M, Sherf M, Mosseri M. USage of chitosan for Femoral (USF) haemostasis after percutaneous procedures: a comparative open label study. EuroIntervention. 2011 Apr;6(9):1104-9. doi: 10.4244/EIJV6I9A192. PMID 21518684
- [Background] Ferretti L, Qiu X, Villalta J, Lin G. Efficacy of BloodSTOP iX, surgicel, and gelfoam in rat models of active bleeding from partial nephrectomy and aortic needle injury. Urology. 2012 Nov;80(5):1161.e1-6. doi: 10.1016/j.urology.2012.06.048. Epub 2012 Aug 22. PMID 22921708
- [Background] Rathore S, Stables RH, Pauriah M, Hakeem A, Mills JD, Palmer ND, Perry RA, Morris JL. A randomized comparison of TR band and radistop hemostatic compression devices after transradial coronary intervention. Catheter Cardiovasc Interv. 2010 Nov 1;76(5):660-7. doi: 10.1002/ccd.22615. PMID 20506228
- [Background] Cong X, Huang Z, Wu J, Wang J, Wen F, Fang L, Fan M, Liang C. Randomized Comparison of 3 Hemostasis Techniques After Transradial Coronary Intervention. J Cardiovasc Nurs. 2016 Sep-Oct;31(5):445-51. doi: 10.1097/JCN.0000000000000268. PMID 26002786
- [Background] Dai N, Xu DC, Hou L, Peng WH, Wei YD, Xu YW. A comparison of 2 devices for radial artery hemostasis after transradial coronary intervention. J Cardiovasc Nurs. 2015 May-Jun;30(3):192-6. doi: 10.1097/JCN.0000000000000115. PMID 24496325
- [Background] Choi EY, Ko YG, Kim JB, Rhee J, Park S, Choi D, Jang Y, Shim WH, Cho SY. Hemostatic efficacy of hydrophilic wound dressing after transradial catheterization. J Invasive Cardiol. 2005 Sep;17(9):459-62. PMID 16145231
- [Derived] Kang SH, Han D, Kim S, Yoon CH, Park JJ, Suh JW, Cho YS, Youn TJ, Chae IH. Hemostasis pad combined with compression device after transradial coronary procedures: A randomized controlled trial. PLoS One. 2017 Jul 24;12(7):e0181099. doi: 10.1371/journal.pone.0181099. eCollection 2017. PMID 28742134